CLINICAL TRIAL: NCT03164954
Title: Étude Observationnelle Prospective d'Une Alerte Douleur informatisée Automatique Par Les Applications Informatiques hospitalières Des HUG Pour prédire l'Apparition de Douleurs Chroniques Post opératoires
Brief Title: Observational Study of an Automatic Detection of Patients at Risk of Chronic Postoperative Pain ("Alerte Douleur")
Acronym: ALDO
Status: Terminated | Type: Observational
Why Stopped: no recruitement possible for >12 months due to highly reduced surgical activity because of the COVID pandemic, all elective surgery was transferred to private hospitals for several months
Sponsor: Benno Rehberg-Klug (Other)
Responsible Party: Sponsor-Investigator, Benno Rehberg-Klug, médecin adjoint agrégé, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: ALDO
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: automatic risk detection — automatic alert of the risk for CPSP, triggered by one of the following entries in the hospital information system: psychological risk factors (depression, anxiety, PTSD, catastrophizing, high pain anticipation), chronic use of benzodiazepines or opioids, intense postoperative pain or need of large opioid doses in the recovery room

SUMMARY:
Following surgery, some but not all patients develop persistent (or chronic) postoperative pain CPSP. Several risk factors for this persistent pain have been confirmed in previous studies, but neither surgeons nor anesthesiologists have or take the time to systematically screen patients for this risk. However, hospital information systems often contain the data already, entered during preoperative consultations (e.g. chronic opioid medication) or obtained during the postoperative period (e.g. pain scores).

Here the investigators test an automatic detection algorithm which alerts the analgesia team when a patient at risk of CPSP is or has been operated.

DETAILED DESCRIPTION:
The primary aim of the study is to confirm that the sensitivity of the automatic alert is at least 80%, i.e. that 80% of patients with the primary outcome had an automatic alert.

The secondary aim of the study is to develop an algorithm (combination of risk factors) with which the specificity of the alert can be improved.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* elective surgery
* perioperative use of the hospital information system
* surgery of the following types: endoprosthesis of the knee or shoulder, amputation other than toe or finger, spinal surgery, cardio-thoracic thoracotomy, laparotomy, inguinal hernia repair, breast surgery

Exclusion Criteria:

* inability to read and understand the consent form or the questionnaires
* emergency surgery
* having already participated in the study for another surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elective surgery
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
CPSP at 6 months | 6 months
  mean pain intensity in the "brief pain inventory" of at least 3/10

SECONDARY OUTCOMES:
CPSP at 12 months | 12 months
  mean pain intensity in the "brief pain inventory" of at least 3/10
clinically significant pain at 6/12 months | 6/12 months
  either a pain intensity of >=3 at rest or >=5 on movement or use of analgesics
neuropathic pain at 6/12 months | 6/12 months
  mean pain intensity in the "brief pain inventory" of at least 3/10 AND a DN4 score of at least 4
acute postoperative pain | 24h postoperative
  mean pain score and highest pain score in the first 24h postoperative on a 0-10 verbal numeric rating scale
pain-related functional deficit at 6/12 months | 6/12 months
  pain interference scales of the brief pain inventory, number of days not working
persistent opioid use | 6/12 months
  patient reported use of tramadol (yes/no) or use of strong opioids (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Bourezg, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
part of the data will be entered into the international Pain-Out database